CLINICAL TRIAL: NCT00215267
Title: The Effect of One Versus Two Praziquantel Treatments on Schistosoma Mansoni Morbidity and re-Infection Along Lake Victoria in Uganda
Brief Title: The Effect of Praziquantel Treatment on Schistosoma Mansoni Morbidity and re-Infection Along Lake Victoria, Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DBL -Institute for Health Research and Development (Other)
Collaborators: Ministry of Health, Uganda (Other Government)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS02310105
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Schistosomiasis; Malaria
Keywords: Schistosoma mansoni; hepatosplenomegaly; malaria; Uganda
MeSH Terms: conditions — Schistosomiasis; Malaria | interventions — Praziquantel

INTERVENTIONS:
Drug: praziquantel

SUMMARY:
The overall objective of the project is to contribute to an increased knowledge about the effect of praziquantel on schistosomiasis related morbidity and re-infection level among communities living along Lake Victoria in Mayuge district, Uganda with the overall aim of improving the strategies for morbidity control.

The study will be carried out in a high transmission area along Lake Victoria, in Mayuge district. It will be a randomised intervention study, comparing a single praziquantel treatment (40mg/kg) with two standard doses administered two weeks apart.

DETAILED DESCRIPTION:
In Uganda, schistosomiasis affects approximately 10% of the population and transmission takes place along all large water bodies (rivers and lakes).

Morbidity control should aim at increasing the length of time before morbidity reappears and decrease the time during which morbidity regresses in a situation with continued transmission and re-infection. It is proposed to test this by comparing the standard treatment with a double treatment (2 x 40 mg/kg) two weeks apart.

The overall objective of the project is to contribute to an increased knowledge about the effect of praziquantel on schistosomiasis related morbidity and re-infection level among communities living along Lake Victoria in Mayuge district, Uganda with the overall aim of improving the strategies for morbidity control.

The study will be carried out in a high transmission area along Lake Victoria, in Mayuge district. It will be a randomised intervention study, comparing a single praziquantel treatment (40mg/kg) with two standard doses administered two weeks apart. Two groups of participants, with 270 people in each, will be randomly selected and randomly assigned to the two treatment regimens. Three consecutive stool samples will be from the cohort and blood samples for malaria will be examined. Clinical and ultrasonographic examinations will be performed. After all the examinations, the whole cohort will be treated with a single standard dose of praziquantel and albendazole. Two weeks later all members of one of the groups will receive another standard dose of praziquantel. Follow-up examinations will be performed 8 weeks, 6 months and two years later.

ELIGIBILITY:
Inclusion Criteria:

* age > 7 years Residence in project village

Exclusion Criteria:

* persons treated with praziquantel within 2 weeks before recruitment

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-09 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
cure rates
re-infection
pathology regression

CONTACTS AND LOCATIONS:
Overall Officials: Edridah M Tukahebwa, Msc, Principal Investigator — Ministry of Health, Uganda
Locations (1):
- Musoli village, Busuyi Parish, Mayuge District, Uganda

REFERENCES:
- [Derived] Kildemoes AO, Vennervald BJ, Tukahebwa EM, Kabatereine NB, Magnussen P, de Dood CJ, Deelder AM, Wilson S, van Dam GJ. Rapid clearance of Schistosoma mansoni circulating cathodic antigen after treatment shown by urine strip tests in a Ugandan fishing community - Relevance for monitoring treatment efficacy and re-infection. PLoS Negl Trop Dis. 2017 Nov 13;11(11):e0006054. doi: 10.1371/journal.pntd.0006054. eCollection 2017 Nov. PMID 29131820
- [Derived] Tukahebwa EM, Vennervald BJ, Nuwaha F, Kabatereine NB, Magnussen P. Comparative efficacy of one versus two doses of praziquantel on cure rate of Schistosoma mansoni infection and re-infection in Mayuge District, Uganda. Trans R Soc Trop Med Hyg. 2013 Jun;107(6):397-404. doi: 10.1093/trstmh/trt024. Epub 2013 Apr 17. PMID 23596262
- See also: Related Info — http://www.dblnet.dk